CLINICAL TRIAL: NCT01849497
Title: A Multi-center, Randomized Study in Subjects With Primary Hypercholesterolemia or Mixed Dyslipidemia to Assess Subjects' Ability to Administer a Full Dose of Evolocumab (AMG 145) in Home-use, Using Either a Prefilled Syringe or a Prefilled Autoinjector/Pen
Brief Title: Study to Assess In-home Use of Evolocumab (AMG 145) Using a Prefilled Syringe or a Prefilled Autoinjector/Pen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120348
Record Dates: First submitted 2013-04-01; First posted 2013-05-08 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia
Keywords: LDL-C, triglycerides, high cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evolocumab PFS (Experimental): Participants received evolocumab 140 mg every 2 weeks for 4 weeks (Day 1, Week 2, and Week 4) subcutaneously using a prefilled syringe (PFS). Participants self-administered evolocumab in the clinic on Day 1 under supervision and then self-administered in a home setting at Weeks 2 and 4.
  Interventions: Biological: Evolocumab Pre-filled Syringe
- Evolocumab AI/pen (Experimental): Participants received evolocumab 140 mg every 2 weeks for 4 weeks (Day 1, Week 2, and Week 4) subcutaneously using a prefilled autoinjector/pen (AI/pen). Participants self-administered evolocumab in the clinic on Day 1 under supervision and then self-administered in a home setting at Weeks 2 and 4.
  Interventions: Biological: Evolocumab AI/pen

INTERVENTIONS:
Biological: Evolocumab Pre-filled Syringe — Evolocumab subcutaneous injection via a single use, disposable pre-filled syringe.
  Other Names: AMG 145; Repatha
  Arms: Evolocumab PFS
Biological: Evolocumab AI/pen — Evolocumab subcutaneous injection via a handheld mechanical (spring-based) autoinjector/pen.
  Other Names: AMG 145; Repatha
  Arms: Evolocumab AI/pen

SUMMARY:
The primary objective of this study was to assess users' ability to administer a full dose of evolocumab in home-use using either a pre-filled syringe or autoinjector/pen.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-C at screening > 85 mg/dL
* Fasting triglycerides less than or equal to 400 mg/dL (4.5 mmol/L) Exclusion Criteria:
* New York Heart Association (NYHA) III or IV heart failure
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension
* Type 1 diabetes or poorly controlled type 2 diabetes
* Uncontrolled hypothyroidism or hyperthyroidism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2013-04-18 (Actual); Primary Completion 2013-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (24):
- United States (20):
  - Research Site, Encino, California
  - Research Site, Thousand Oaks, California
  - Research Site, Ventura, California
  - Research Site, Westlake Village, California
  - Research Site, Miami, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Hammond, Indiana
  - Research Site, Auburn, Maine
  - Research Site, Manlius, New York
  - Research Site, Syracuse, New York
  - Research Site, Cadiz, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Hillsboro, Oregon
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Lansdale, Pennsylvania
  - Research Site, Rapid City, South Dakota
  - Research Site, Jackson, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Canada (4):
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Woodstock, Ontario
  - Research Site, Pointe-Claire, Quebec

REFERENCES:
- [Background] Boccara F, Dent R, Ruilope L, Valensi P. Practical Considerations for the Use of Subcutaneous Treatment in the Management of Dyslipidaemia. Adv Ther. 2017 Aug;34(8):1876-1896. doi: 10.1007/s12325-017-0586-8. Epub 2017 Jul 17. PMID 28717862
- [Background] Toth PP, Descamps O, Genest J, Sattar N, Preiss D, Dent R, Djedjos C, Wu Y, Geller M, Uhart M, Somaratne R, Wasserman SM; PROFICIO Investigators. Pooled Safety Analysis of Evolocumab in Over 6000 Patients From Double-Blind and Open-Label Extension Studies. Circulation. 2017 May 9;135(19):1819-1831. doi: 10.1161/CIRCULATIONAHA.116.025233. Epub 2017 Mar 1. PMID 28249876
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Derived] Dent R, Joshi R, Stephen Djedjos C, Legg J, Elliott M, Geller M, Meyer D, Somaratne R, Recknor C, Weiss R. Evolocumab lowers LDL-C safely and effectively when self-administered in the at-home setting. Springerplus. 2016 Mar 9;5:300. doi: 10.1186/s40064-016-1892-3. eCollection 2016. PMID 27066336
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were men and women ≥ 18 and ≤ 80 years of age with fasting low-density lipoprotein cholesterol (LDL-C) ≥ 85 mg/dL, fasting triglycerides ≤ 400 mg/dL and on a stable dose of a statin with or without ezetimibe for at least 4 weeks.
  The first patient enrolled on 18 April 2013 and last patient enrolled on 05 August 2013.
Pre-assignment Details: Randomization was stratified on the basis of screening LDL-C concentration (< 130 mg/dL [3.4 mmol/L] or ≥ 130 mg/dL). Participants were trained by study site staff to prepare and self-administer the study drug.
Period: Overall Study
Arm/Group | Evolocumab PFS | Evolocumab AI/Pen
Started | 75 | 74
Received Treatment | 75 | 74
Completed | 74 | 70
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Sponsor Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (all randomized participants who received at least 1 dose of study drug).
Groups:
- Evolocumab PFS: Participants received evolocumab 140 mg every 2 weeks for 4 weeks (Day 1, Week 2, and Week 4) subcutaneously using a prefilled syringe (PFS).
- Evolocumab AI/Pen: Participants received evolocumab 140 mg every 2 weeks for 4 weeks (Day 1, Week 2, and Week 4) subcutaneously using a prefilled autoinjector/pen (AI/pen).
- Total: Total of all reporting groups
Arm/Group | Evolocumab PFS | Evolocumab AI/Pen | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (11.1) | 60.6 (9.6) | 60.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 26 | 62
  Male | 39 | 48 | 87
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 7 | 9
  Black or African American | 11 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 62 | 58 | 120
  Missing | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 66 | 68 | 134
Stratification Factor: LDL-C Level [Number; unit: participants]
  < 130 mg/dL | 56 | 56 | 112
  ≥ 130 mg/dL | 19 | 18 | 37
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] | 116.9 (25.0) | 118.1 (28.7) | 117.5 (26.8)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Full Administration of Evolocumab at Both Weeks 2 and 4
Description: Self-administration of evolocumab was assessed by a telephone interview at Weeks 2 and 4. Each participant was asked about all attempted injection(s) and if the injection was administered in part, full, or none at all.
Time Frame: Week 2 and Week 4
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Evolocumab PFS | Evolocumab AI/Pen
Number analyzed (Participants) | 75 | 74
percentage of participants | 96.0 [88.9 to 98.6] | 89.2 [80.1 to 94.4]
Statistical Analysis 1: Comparison: Evolocumab PFS vs Evolocumab AI/Pen; Test type: Superiority or Other; Treatment Difference = -6.8, 95% CI 2-sided [-16.3 to 2.0]

2. Secondary Outcome: Percent Change From Baseline in LDL-C at Week 6
Time Frame: Baseline and Week 6
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Evolocumab PFS | Evolocumab AI/Pen
Number analyzed (Participants) | 75 | 74
percent change | -59.74 (2.57) | -63.43 (2.67)
Statistical Analysis 1: Comparison: Evolocumab PFS vs Evolocumab AI/Pen; Test type: Superiority or Other; LS Mean Treatment Difference = -3.70, 95% CI 2-sided [-10.38 to 2.99], Standard Error of Mean 3.38

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 28 days after last study drug administration (up to 8 weeks)
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Evolocumab PFS | Evolocumab AI/Pen
Serious Adverse Events (participants affected / at risk) | 3/75 | 2/74
Other Adverse Events (participants affected / at risk) | 4/75 | 2/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab PFS (N=75) | Evolocumab AI/Pen (N=74)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Glomerulonephritis minimal lesion (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab PFS (N=75) | Evolocumab AI/Pen (N=74)
Headache (Nervous system disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.